CLINICAL TRIAL: NCT03018002
Title: Intervention for Sustained Testing and Retention Among HIV-infected Patients
Acronym: iSTAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Echezona Ezeanolue, Professor of Public Health and Pediatrics, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 845695-4; R01HD087994-01 (NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: HIV
Keywords: HIV, PMTCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): HIV-infected participants identified from the churches randomized to CG will be referred to PEPFAR-supported HIV clinics that provide comprehensive care including counseling, laboratory testing, ART and ongoing support during treatment as the standard of care. The study team will not be involved in their care beyond data collection.
- iSTAR (Experimental): HIV-infected participants identified from the churches clustered within the randomized health facilities will receive interventions from the study team.
  Interventions: Other: iSTAR

INTERVENTIONS:
Other: iSTAR — Each component of the iSTAR intervention targets a specific point along the HIV continuum: confidential, onsite integrated laboratory tests during baby showers targets HIV diagnosis (b) church-based Health Advisors (CHAs) trained in motivational interviewing and quality improvement skills as promotoras target linkage, engagement and adherence by providing counseling and other support to HIV-infected women and children (c) integrated network of community and clinic case management targets reduction in loss to follow-up.
  CHAs will support participants during the study period by being available to accompany them to clinic visits, review laboratory results and medications after clinic visits. They will be available to speak with them at intervals to see how they are doing either by phone or through home visits as they prefer. At each follow-up study visit, the trained CHA will review and collect data on participants' clinic visits, treatment, and laboratory results.
  Arms: iSTAR

SUMMARY:
The purpose of this study is to evaluate the comparative effectiveness of a congregation, clinic and integrated case management-based intervention for sustainable testing and retention on linkage to care, engagement, retention and viral load suppression of women and children infected with HIV.

DETAILED DESCRIPTION:
Using a two-arm cluster randomized design, our proposed study will evaluate the comparative effectiveness of iSTAR, a community-based social network intervention that combines trained church-based Health Advisors and clinic-based staff and uses motivational interview skills and clinic- quality improvement approaches (Intervention Group; IG) versus a clinic-based approach (Control group; CG) on linkage, engagement, retention and viral suppression among HIV-infected women and children. Eighteen health facilities in identified local government areas in Benue state, north-central Nigeria will be randomly assigned to either the IG (N=9 health facilities) or the CG (N=9 health facilities). A total of 10,000 pregnant women will be screened and 400 HIV-infected participants will be enrolled over a 24-month period. The primary outcome will be the difference in the rate of linkage and engagement between the groups. The secondary outcome will be the difference in rate of retention and viral suppression among participants. Additionally, we will conduct network, mediation/moderation analysis to examine the roles of intermediate variables such as health team cohesion, turnovers, attitudes, leadership and dynamic adaptation on iSTAR implementation and sustainment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected pregnant women identified during baby showers programs at participating worship centers.

Exclusion Criteria:

* HIV-infected women already on treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Linkage in care | 1 month
  Linkage in care is defined as the percentage of participants with at least one HIV medical care visit following HIV diagnosis.
Retention in care | 12 months
  Retention is defined as the percentages of participants with two or more documented viral load measurement during the 12 months following enrollment.

SECONDARY OUTCOMES:
ART Initiation | 1 month
  The secondary outcome is engagement in care defined as the percentage of participants initiated on ART at 1 month following enrollment.
Viral Suppression | 12 months
  Viral suppression is defined as the percentage of participants whose most recent two viral load are <20 copies/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Caritas Foundation, Makurdi, Benue State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezeanolue EE, Obiefune MC, Yang W, Obaro SK, Ezeanolue CO, Ogedegbe GG. Comparative effectiveness of congregation- versus clinic-based approach to prevention of mother-to-child HIV transmission: study protocol for a cluster randomized controlled trial. Implement Sci. 2013 Jun 8;8:62. doi: 10.1186/1748-5908-8-62. PMID 23758933